CLINICAL TRIAL: NCT02490579
Title: Effectiveness of Video Messaging About Diet, Exercise and Weight Gain in Pregnancy in Regional and National Samples
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Michelle H. Moniz, Assistant Professor, University of Michigan
Other Study IDs: HUM00101358
Record Dates: First submitted 2015-06-29; First posted 2015-07-07 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy; Weight Gain
Keywords: video messaging; exercise; diet; weight gain; pregnancy
MeSH Terms: conditions — Weight Gain; Motor Activity | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Facebook Survey Group: During June, 2015, approximately 1200 women will be recruited through Facebook advertisements targeted at English-speaking women age 18-50 years living in the United States. Advertisements will contain 3 key features: an image, a caption, and "ad copy" followed by a link to the survey website. Individuals who click on the study link in the advertisement will be redirected to the study's Qualtrics web page where they will take a 15 web-page, multiple choice survey developed by the research team. The survey covers these domains: reaction to video, understanding of core message, self-efficacy around lifestyle behaviors, attitudes, beliefs and intentions regarding vaccination during pregnancy, key health information sources during pregnancy, and demographics.
  Interventions: Behavioral: Responses to Brief Video Messages (Facebook)
- Clinical Survey Group: During June-August, 2015, approximately 500 women will be recruited at routine obstetric visits to the University of Michigan's outpatient clinics. Women who check in for an Ob appointment will be offered the opportunity to participate in an anonymous online survey. Individuals who express interest in participating will be provided with a laptop and headphones and directed to the survey Qualtrics site where they will take a 15 web-page, multiple choice survey developed by the research team. The survey covers these domains: reaction to video, understanding of core message, self-efficacy around lifestyle behaviors, attitudes, beliefs and intentions regarding vaccination during pregnancy, key health information sources during pregnancy, and demographics.
  Interventions: Behavioral: Response to Brief Video Messages (Clinic)
- Social Network Group: Once a pregnant participant completes the survey, she will be asked to provide her email address. If she is willing to do so, Qualtrics will automatically send her an email containing a weblink to the survey for her social network. She can then provide this link to 1 or 2 social network members that she feels influence her health behaviors during pregnancy. These members are asked similar questions about their response to the video, as well as some additional questions about how they advise their pregnant person about different health topics. It is necessary to provide a unique weblink to her, so that the survey responses from the pregnant woman and her unique social network members can be linked.
  Interventions: Behavioral: Response to Brief Video Messages (Social Network)

INTERVENTIONS:
Behavioral: Responses to Brief Video Messages (Facebook) — Participants view 1 of 6 brief video messages about health in pregnancy, then answer survey questions that will assess their a) acceptability, b) understanding of core messages, and c) self-efficacy about healthy eating, exercise and weight gain during pregnancy.
  Groups: Facebook Survey Group
Behavioral: Response to Brief Video Messages (Clinic) — Participants view 1 of 6 brief video messages about health in pregnancy, then answer survey questions that will assess their a) acceptability, b) understanding of core messages, and c) who in her social network she turns to for non-clinical health advice and what kinds of advice she gotten in the past.
  Groups: Clinical Survey Group
Behavioral: Response to Brief Video Messages (Social Network) — Participants view 1 of 6 brief video messages about health in pregnancy, then answer survey questions that will assess their a) acceptability, b) understanding of core messages, and c) how they advise their pregnant friend about different health topics.
  Groups: Social Network Group

SUMMARY:
The primary purpose of this study is to assess the responses of pregnant women and their social network to six videos about health in pregnancy. Our goal is to assess a) acceptability and b) understanding of core messages about healthy eating, exercise and weight gain during pregnancy. We will also assess c) non-clinical sources of health information during pregnancy.

DETAILED DESCRIPTION:
Many women engage in suboptimal lifestyle behaviors during pregnancy. Many women do not realize that unhealthy diet, exercise and weight gain behaviors can be dangerous for their pregnancy and have harmful long-term consequences for their baby. There is great need for strategies to promote accurate knowledge about healthy behaviors during pregnancy. The purpose of this study is to assess responses to a brief (<1minute) video about healthy behaviors during pregnancy. The study sample will include pregnant women and members of their social network. Participants will be asked to watch a brief video and complete an anonymous online survey measuring their response to the video, and their basic demographics. The surveys will also assess how family and friends impact pregnant women's health behaviors. Online surveys are entirely anonymous. We will recruit pregnant participants from two sources: the University of Michigan Health System's prenatal clinics and a social media website (Facebook).

ELIGIBILITY:
Inclusion Criteria:

* Women
* Currently Pregnant
* Age 18 or over
* English-speaking

Exclusion Criteria:

* Deny being currently pregnant
* Do not identify as living in the US and aged 18 years or older
* Report having previously participated in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women recruited via either the social media, clinical, or online approach will be eligible for participation if they are aged 18 years and older, pregnant, and English-speaking. Women will be excluded if they deny being currently pregnant, do not identify as living in the US and aged 18 years or older, or if they report having previously participated in the study. The Qualtrics survey will automatically conclude if potential participants provide answers to screening questions that deem them ineligible. Participants will not be excluded based on racial-ethnic groups. Males will be excluded, as this is a study involving pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 1670 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Composite acceptability score (continuous variable) | 15 minutes
  Participants will be asked questions about their reaction to the video.
Understanding of core messages (free text item; categorical items) | 15 minutes
  Trained research assistants will review answers to questions regarding diet, exercise and weight gain in pregnancy to determine whether individuals understood/did not understand the core message.
Self-efficacy (continuous scale; Facebook group only) | 15 minutes
  Participants will answer questions about self-efficacy regarding weight gain, exercise and diet.
Sources of information about health during pregnancy (categorical variable; clinic and social network groups only) | 15 minutes
  Participants will answer questions about what sources of health information are provided by social network contacts during pregnancy.
Content of health information from interpersonal sources during pregnancy (free text variable; clinic and social network groups only) | 15 minutes
  Trained research assistants will review answers to questions about the types of health information and advice are provided by social network contacts during pregnancy.
Perceived impact of interpersonal health advice on health behaviors during pregnancy (categorical and free text variables; clinic and social network groups only) | 15 minutes
  Participants answer questions about the impact the health information and advice they receive from social network contacts during pregnancy has on their behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle H. Moniz, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No